CLINICAL TRIAL: NCT06780709
Title: Impact of a Structured Wellness Behavioral Intervention on Quality of Life in NMOSD
Acronym: NMOSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Sammita Satyanarayan, Assistant Professor, Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-23-01257; ISRA# 370464 (Other Grant/Funding Number: Amgen)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neuromyelitis Optica Spectrum Disorder (NMOSD)
Keywords: NMOSD; Wellness; Diet; Physical Therapy; Social Work; Comprehensive
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Health Promotion; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two assigned arms of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Start (Experimental): Participants will begin wellness program services and behavioral interventions immediately after randomization
  Interventions: Behavioral: Wellness Program and Behavioral Counseling
- Delayed Start (Other): Participants will experience a 6-month delay in receiving wellness program services and behavioral interventions.
  Interventions: Behavioral: Wellness Program and Behavioral Counseling

INTERVENTIONS:
Behavioral: Wellness Program and Behavioral Counseling — The comprehensive wellness evaluation will include initial assessments by dietician, social worker, physical therapist, nurse practitioner, and a behavioral neuropsychologist. Each provider will conduct an initial evaluation at baseline to identify areas of need and patient driven goals, as well as follow-up evaluations to evaluate implementation of changes and barriers to change.

SUMMARY:
This project aims to study whether a structured wellness program intervention can improve quality of life among people living with Neuromyelitis Optica Spectrum Disorder (NMOSD). This pilot will test a multi-modal wellness program tailored to NMOSD patients that includes services from physical therapists, dietitians, social workers, nurse practitioners and cognitive therapists. The trial will be designed as a randomized controlled trial, randomizing patients to immediately starting the program as well as a 6 month delayed start. The intervention would leverage an existing clinical comprehensive MS wellness program at the Corinne Dickinson for Multiple Sclerosis (MS) at Mount Sinai Medical Center. The primary endpoint of this study would be evaluating quality of life, as assessed by MS-Quality of Life -54.

DETAILED DESCRIPTION:
This pilot will aim to recruit 20 patients. Participants will be randomized into one of two arms: the trial group will begin wellness program services and behavioral interventions immediately; the control group will participate in other educational activities, and begin wellness program services and behavioral interventions 6 months after randomization. The wellness intervention will include dietary, physical therapy, social work, and nurse practitioner evaluations, as well as behavioral counseling to implement recommendations. All participants will complete assessments, with patient-reported outcome surveys and objective assessments at baseline, 12 weeks, and 6 months for the core study. Participants will also be offered the option of continuing into a one year extension study, wherein one additional wellness intervention and bimonthly behavioral counseling sessions will be offered until 12 months on study. Study assessments will be completed at 12 months and 18 months to assess sustainability of the program. Assessments will include subjective reports of quality of life as pertaining to living with their disease, mobility, vision, exercise, diet, as well as objective measures of motor and vision function.

ELIGIBILITY:
Inclusion criteria:

* Adults (age ≥18) with NMOSD diagnosed with 2015 NMOSD clinical criteria.
* All EDSS scores will be considered in order to make the intervention accessible to all patients regardless of disability.
* All patients regardless of treatment type will be considered.

Exclusion criteria:

* Age<18
* Inability to voluntarily provide consent for study participation
* Inability to participate in study evaluation and/or endpoint measures, or participation in another concurrent randomized controlled trial or wellness based intervention.
* Any patients with a relapse within 30 days of randomization or any patients with medical restrictions on physical activity will be excluded.
* Any patients who begin stimulants and/or dalfampridine between enrollment and randomization will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Quality of Life (MSQOL-54) Score | at baseline, 3 months, at 6 months, at 12 months for extension study, at 18 months for extension study
  The MSQOL-54 is a 54-item comprehensive patient-reported questionnaire for individuals with MS.
  MSQOL-54 yields two main composite scores calculated using weighted averages of relevant areas: Physical Health Composite (PHC) - the physical function, health perceptions, energy/fatigue, role limitations- physical, pain, sexual function, social function, health distress scales. The Mental Health Composite (MHC) - the health distress, overall quality of life, emotional wellbeing, role limitations- emotional, cognitive function scales.
  Each composite scores range from 0-100, with total scale range from 0-100. Higher scores indicating better perceived health and quality of life. Lower scores suggest poorer quality of life impacted by MS. MSQOL-54 evaluates how MS affects various aspects of a patient's life and well-being, providing valuable insights into the patient's overall health status and the impact of MS on their daily functioning.

SECONDARY OUTCOMES:
Impact of vision impairment (IVI) Score | at baseline, 3 months, at 6 months, at 12 months for extension study, at 18 months for extension study
  The Impact of Vision Impairment (IVI) is a 32-item patient-reported instrument measuring vision impairment's effect on quality of life and daily activities. The questionnaire assesses five domain subscales: Leisure and Work, Social and Consumer Interaction, Household and Personal Care, Mobility, and Emotional Reaction to Vision Loss. Items use a 6-point Likert scale (0: Not at all, 1: Hardly at all, 2: A little, 3: A fair amount, 4: A lot, 5: Can't do because of eyesight). Domain subscale scores are calculated as the mean of items within each domain, and the total score is the mean of all items. Subscales range from 0-5, with total scale range from 0-5. Lower scores indicating better vision-related quality of life. A decrease in scores represents improvement over time.
Neuro-Quality of Life (Neuro-QOL) Score | at baseline, 3 months, at 6 months, at 12 months for extension study, at 18 months for extension study
  Neuro QOL (quality of life) subscales indicating upper extremity function, lower extremity function, executive function, ability to participate in social roles/activities, satisfaction with social roles and activities) will be assessed. Scores are assessed and compared to normative data, with a T score generated. T distributions assume a mean of 50, and the standard deviation is set to 10 units. A higher T score value indicates a greater deviation from normal functioning.
The Godin Leisure Time and Exercise (GLTEQ) Score | at baseline, 3 months, at 6 months, at 12 months for extension study, at 18 months for extension study
  The GLTEQ is a patient reported scale assessing patient reported frequency of exercise in a typical 7-day period during their free time. Total Scale is weighted to calculate a composite score from 0-99, with a higher score indicating a more active lifestyle.
Mediterranean Diet Compliance Scale (MEDAS) | at baseline, 3 months, at 6 months, at 12 months for extension study, at 18 months for extension study
  MEDAS questionnaire is a self-reported recall of food consumption. This is a 14-item questionnaire, with each item being scored as a 0 or 1 indicating consumption of the specified category of food, with a total scale range of 0-14. A higher score indicates a higher alignment with a mediterranean based diet.

CONTACTS AND LOCATIONS:
Overall Officials: Sammita Satyanarayan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Corinne Goldsmith Dickinson Center for MS at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Dataset includes sensitive data such as substance use (from dietary surveys) and mental health status.